CLINICAL TRIAL: NCT03575546
Title: Clinical and Functional Outcome of the Gemini SL Fixed Bearing at Midterm Follow-up
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Waldemar Link GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: KP05A
Record Dates: First submitted 2018-06-15; First posted 2018-07-02 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, multicenter case series with a prospective follow-up to confirm the safety and performance of the Gemini SL Fixed Bearing knee prosthesis in midterm follow-up under routine conditions. Primary outcome of the study is the 5-year survival rate of the Gemini SL Fixed Bearing knee prosthesis with revision for any reason as the end point.

DETAILED DESCRIPTION:
Sufficient data (e.g. biomechanical tests, biocompatibility, vigilance data and results of risk management, clinical data of comparable devices) are available for assessing the safety and performance of the Gemini SL knee prosthesis system. Unfortunately, no data are available for the Gemini SL Fixed Bearing knee prosthesis. As one part of the post market surveillance (PMS) system of the sponsor, the clinical outcome of the Gemini SL Fixed Bearing knee prosthesis in the midterm follow-up shall be evaluated. Therefore patients who received a Gemini Sl Fixed bearing knee prosthesis 3 years ago are invited to participate in follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of a Gemini SL Fixed Bearing knee prostheses 3 years ago
* Age between 18 and 75 years at the time of implantation

Exclusion Criteria:

* Body Mass Index (BMI) > 40 kg/m² at the time of implantation
* Comorbidities and known medical circumstances which would affect the clinical functional outcome after implantation of the knee prosthesis (e.g. neurological or musculoskeletal diseases) at the time of implantation
* Prisoner

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients received a Gemini SL Fixed Bearing knee prosthesis in the study sites 3 years ago are possible participants of the study. Hospital charts will be screened in order to identify these candidates. The patients will be followed up at 3-year interval.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Survival rate of the Gemini SL Fixed Bearing knee prosthesis with revision for any reason as the end point | 5 years
  Revision for any reason is defined as removal, replacement or adding of any implant components, except subsequent implantation or replacement of the patella surface or the polyethylene plateau.

SECONDARY OUTCOMES:
Survival rate of the Gemini SL Fixed Bearing knee prosthesis with revision for any reason as the end point | 3 years
  Revision for any reason is defined as removal, replacement or adding of any implant components, except subsequent implantation or replacement of the patella surface or the polyethylene plateau.
Evaluation of the functional and clinical outcome of the Gemini SL Fixed Bearing knee prosthesis measured by the Knee Society Score | 3 and 5 year
  Evaluation of KSS Score (Validated Score)
Complication rates | 3 and 5 years
  Number and kind of complications
Subsequent surgical interventions | 3 and 5 years
  Number and kind of subsequent surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Wülker, Principal Investigator — Universitätsklinikum Tübingen für Orthopädie
Locations (3):
- Germany (2):
  - Klinik Oberammergau, Oberammergau
  - Universitätsklinikum Tübingen für Orthopädie, Tübingen
- Hospital central de la Cruz Roja, Madrid, Spain